CLINICAL TRIAL: NCT04691921
Title: Nation-wide Cross-sectional Survey on Current Pharmacological Practices in Severe COVID-19
Brief Title: Current Pharmacological Practices in Severe COVID-19
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Specialist Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: NMCSH
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Current clinical practices of participating physicians — Current clinical practice of participating physicians on choice of pharmacological agents for clinical management of Severe COVID-19

SUMMARY:
The investigators aim to understand the variation in pharmacological therapies for the management of severe coronavirus disease 2019 (COVID-19) in India and compare it to the recent available evidence.

The ongoing pandemic of COVID-19 has proven to be the greatest medical emergency of recent times. The evidence on the therapeutics has evolved significantly in last few months after initial use of re-purposed drugs.

The objective of this study is to understand the current practices in the management of adults severe COVID-19 in India.

DETAILED DESCRIPTION:
The ongoing pandemic of COVID-19 has proven to be the greatest medical emergency of recent times. The response of the medical world to this crisis has been unprecedented. The healthcare workers are caring for patients at the frontline while, scientists and researchers are discovering vaccines or effective treatment in shortest possible duration. The scale and effect of pandemic in India, being second most populous country of the world is enormous. As of December 30, 2020, India has crossed 10 million cases and 148,000 deaths from COVID-19. India has second most number of cases only after United States of America (USA) and with third largest number of deaths. The Ministry of Health and family Welfare (Under Government of India) has given periodical clinical management guidelines, with last updated on July 5, 2020 (version 5).

In adults, severe COVID-19 is defined as presence of any of the following dyspnea, a respiratory rate of 30 or more breaths per minute, a blood oxygen saturation (SpO2) of 93% or less, a ratio of the partial pressure of arterial oxygen to the fraction of inspired oxygen (Pao2:Fio2) of less than 300 mm Hg, or infiltrates in more than 50% of the lung field while Critical COVID-19 is defined as presence of acute respiratory distress syndrome (ARDS), sepsis or septic shock. The mortality in critical COVID-19 is reported to be 25-49% in different studies. The evidence on the therapeutics for COVID-19 has evolved significantly in last few months after initial use of re-purposed drugs. There are no recent guidelines available based on the current evidence for clinical management of COVID-19.

The investigators are planning for nation-wide multicentre cross-sectional survey on understanding participating physicians practices on choice of different pharmacotherapeutic agents available in India as of January 2021.

The objective of this study is to understand the current practices of participating physicians in the management of adult patients with severe COVID-19 in India and to determine future priorities.

ELIGIBILITY:
Inclusion Criteria:

Physicians who are involved in management of adult patients with severe COVID-19 in India

Exclusion Criteria:

Pediatrician Physicians who are not managing severe COVID-19 patients or refused to participate.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians involved in the clinical management of adult severe COVID-19 patients in India.
Sampling Method: Probability Sample
Enrollment: 1055 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Choice and indication of pharmacological agents for management of Severe COVID-19 | two weeks
  Cross-sectional survey will capture the current choice and indication of different pharmacological agents for management of Severe COVID-19 among participating physicians in India

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Nasa, MD EDICM, Principal Investigator — NMC Specialty Hospital
Locations (1):
- Reliance Hospital, Mumbai, Mumbai, Mahrastra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Result] Berlin DA, Gulick RM, Martinez FJ. Severe Covid-19. N Engl J Med. 2020 Dec 17;383(25):2451-2460. doi: 10.1056/NEJMcp2009575. Epub 2020 May 15. No abstract available. PMID 32412710
- See also: Ministry Of Health and Family Welfare, India. Clinical management of COVID-19 — https://www.mohfw.gov.in/pdf/GuidelinesonClinicalManagementofCOVID1912020.pdf